CLINICAL TRIAL: NCT02821715
Title: Safety and Efficacy of THN102 on Sleepiness in Narcoleptic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theranexus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THN102-201; 2015-005035-41 (EudraCT Number)
Record Dates: First submitted 2016-06-23; First posted 2016-07-01 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — Modafinil; Flecainide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Modafinil + placebo (Active Comparator): 3 tablets modafinil 100 mg per day and 3 capsules flecainide placebo per day for 2 weeks
  Interventions: Drug: Active comparator: Modafinil + placebo
- THN102 300/3 (Experimental): 3 tablets modafinil 100 mg per day and 3 capsules flecainide 1 mg per day (THN102 as 300 + 3 mg) for 2 weeks
  Interventions: Drug: THN102 300/3
- THN102 300/27 (Experimental): 3 tablets modafinil 100 mg per day and 3 capsules flecainide 9 mg per day(THN102 as 300 + 27 mg) for 2 weeks
  Interventions: Drug: THN102 300/27

INTERVENTIONS:
Drug: Active comparator: Modafinil + placebo
  Other Names: Modafinil 300 mg; Flecainide Placebo
  Arms: Modafinil + placebo
Drug: THN102 300/3
  Other Names: Modafinil 300 mg; Flecainide 3 mg
  Arms: THN102 300/3
Drug: THN102 300/27
  Other Names: Modafinil 300 mg; Flecainide 27 mg
  Arms: THN102 300/27

SUMMARY:
This Phase 2 study is a 8-site, double-blind, randomised, placebo-controlled, 3-way cross-over trial, involving 3 treatments with Modafinil 300 mg or the combination drug THN102 (Modafinil/Flecainide 300 /3 mg, Modafinil/Flecainide 300 /27 mg).

DETAILED DESCRIPTION:
The 3 double blind periods (2-week) follow a stabilisation period for modafinil at 300 mg/day (open, 2-week) and are followed by a one-week washout period with the same modafinil dose.

ELIGIBILITY:
Main inclusion Criteria:

* Patients with a diagnosis of narcolepsy type 1 (i.e. with cataplexy) or type 2 (without cataplexy) according to the International Classification of Sleep Disorders (ICSD-3) criteria.
* Body mass index >18 kg/m2 and <35 kg/m2.
* Patients treated with modafinil at stable dosage for at least 2 months and still complaining of excessive daily somnolence (EDS) despite the treatment
* Epworth Sleepiness Scale (ESS) score should be ≥ 14/24 during the baseline period.

Main exclusion Criteria:

* Patients with an untreated sleep apnea syndrome (respiratory disorder index > 30/h) or who have any other cause of daytime sleepiness as assessed on patient history.
* Psychiatric and neurological disorders, other than narcolepsy/cataplexy, such as Parkinson's disease, Alzheimer's disease, Huntington's Chorea, multiple sclerosis, moderate or severe psychosis or dementia, bipolar illness, epilepsy, severe clinical anxiety or depression, Beck Depression Inventory ≥ 21 or with suicidal risk (if item > 0), or other problem that in the investigator's opinion would preclude the patient's participation and completion of this trial or comprise reliable representation of subjective symptoms.
* Contraindication to flecainide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Dauvilliers, MD, PhD, Principal Investigator — CHRU Montpellier, France
Locations (8):
- RespiSom, Erpent, Belgium
- France (7):
  - CHU Pellegrin, Bordeaux
  - CHU Dijon Bourgogne, Dijon
  - Hôpital Raymond Poincaré, Garches
  - CHU Grenoble Alpes, Grenoble
  - CHRU Lilles, Lille
  - University Hospital, Montpellier
  - Groupe Hospitalier Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 patients were screened, 51 patients were randomized and 48 started the double-blind treatment period
Pre-assignment Details: Study starts with open-label run in period with modafinil 300 mg/d. 51 patients met study inclusion/exclusion criteria and entered the run-in period, 48 subjects still fulfilled inclusion criteria after run-in and entered the double-blind period.
Groups:
- Sequence 1 : ABC; Sequence 2 : BCA; Sequence 3: CAB; Sequence 4: ACB; Sequence 5: CBA; Sequence 6: BAC: Treatment A : 300 mg modafinil + 0 mg flecainide per day Treatment B : 300 mg modafinil and 3 mg flecainide per day Treatment C: 300 mg modafinil and 27 mg flecainide per day
  Treatment period A, B and C duration = 2 weeks No wash out between each period
Period: Overall Study
Arm/Group | Sequence 1 : ABC | Sequence 2 : BCA | Sequence 3: CAB | Sequence 4: ACB | Sequence 5: CBA | Sequence 6: BAC
Started | 8 | 8 | 8 | 9 | 6 | 9
Completed | 7 | 8 | 8 | 9 | 6 | 9
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Ethnicity data not collected at baseline
Groups:
- All Participants: Participants received either:
  A Modafinil 300mg/d/Flecainide placebo, B Modafinil 300mg/d/Flecainide 3mg/d C Modafinil 300mg/d/Flecainide 27mg/d
Arm/Group | All Participants
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 51 patients were randomised (1 randomized patient never took study medication), Safety set: 50 patients Modified Intent to Treat Set: 48 patients
  Participants
    Female | 24
    Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 4
  France | 47
Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — Score from 0 to 24, high score = severe sleepiness Population: Efficacy population (modified Intent to Treat Population) 48
  units on a scale
    number analyzed (Participants) | 48
    (all) | 17.1 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Epworth Sleepiness Scale (ESS)
Description: Range 0 to 24, low score indicates good outcome
Time Frame: 14 days after the beginning of treatment period
Population: modified Intent To Treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Modafinil + Placebo: 3 tablets modafinil 100 mg per day and 3 capsules flecainide placebo per day for 2 weeks
  Active comparator: Modafinil + placebo
- THN102 300/3: 3 tablets modafinil 100 mg per day and 3 capsules flecainide 1 mg per day (THN102 as 300 + 3 mg) for 2 weeks
  THN102 300/3
- THN102 300/27: 3 tablets modafinil 100 mg per day and 3 capsules flecainide 9 mg per day(THN102 as 300 + 27 mg) for 2 weeks
  THN102 300/27
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 48 | 48 | 48
score on a scale | 14.68 (0.689) | 15.34 (0.695) | 15.34 (0.694)

2. Secondary Outcome: 14-item Fatigue Scale
Description: Fatigue scale is a rating scale completed by the participants at each visit starting from baseline to last visit; 14 questions to be ticked off by "yes" or "No" by the patient. 0 : No fatigue 14 : worst fatigue condition
Time Frame: 14 days after the beginning of treatment period
Population: modified Intent To Treat (mITT)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 47 | 47 | 46
score on a scale | 6.37 (0.545) | 6.94 (0.549) | 7.25 (0.549)

3. Secondary Outcome: Questionnaire EQ-5D (European Quality of Life EQ-5D) (Questionnaire Part)
Description: EQ-5D is a quality of life questionnaire filled in by the participants from screening to the last visit (all visits).
  The EQ-5D assesses the status on the day of visit and not over the past week. It has two parts:
  The first part is a descriptive system that assesses five distinct health states/dimensions: Mobility (MO), Self-care (SC), Usual activities (UA), Pain/discomfort, Anxiety/depression (AD). A higher score signifies a higher number of symptoms present.
  The second part is a 100 mm VAS (EQ-VAS). An increase in VAS indicates an improvement in health state.
Time Frame: 14 days after the beginning of the screening
Population: mITT
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 47 | 46 | 46
score on a scale | 0.86 (0.358) | 1.16 (0.189) | 1.24 (0.258)

4. Secondary Outcome: Patient Global Impression of Change (PGI-C)
Description: PGI-C is a scale completed by the participants starting from screening to last Last visit (all the visits).
  Participants have to chose 1 condition among 7 : Very much improved/ Much improved/ Minimally improved/ No change/ Minimally worse/ Much worse/ Very much worse.
  1 is the best score (very much improved) 7 is the worse score (very much worse)
Time Frame: 14 days after the beginning of treatment period
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 46 | 46 | 46
Participants
  Very much improved | 2 | 1 | 0
  Much improved | 10 | 7 | 9
  Minimally improved | 16 | 15 | 10
  No change | 10 | 12 | 17
  Minimally worse | 8 | 7 | 8
  Much worse | 0 | 3 | 1
  Very much worse | 0 | 1 | 1

5. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Global Impression
Description: CGI-C (change from baseline) is a scale completed by the investigator at V3, V4 , V5 and V6 for global impression the investigator or his/her designee has to score 3 items : global impression/ sleepiness and Cataplexy.
  For each item the investigator or his/her designee has to chose 1 condition among 7 : Very much improved/ Much improved/ Minimally improved/ No change/ Minimally worse/ Much worse/ Very much worse.
  1 is the best score (very much improved) 7 is the worse score (very much worse)
Time Frame: 14 days after the end of treatment period I
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 47 | 47 | 47
Participants
  Very much improved | 3 | 1 | 0
  Much improved | 7 | 10 | 8
  Minimally improved | 18 | 9 | 13
  no change | 14 | 21 | 21
  Minimally worse | 4 | 3 | 5
  Much worse | 1 | 2 | 0
  Very much worse | 0 | 1 | 0

6. Secondary Outcome: Beck Depression Inventory (BDI)
Description: Beck Depression Inventory (BDI) evaluation for depressive symptoms (including suicidal thoughts). The scale is completed by the participants from baseline, to last visit (all except screening visit). The questionnaire contains 21 items. Each must be scored from 0 to 3, minimum score = 0, maximum score = 63. A high score indicates increased severity of depression.
Time Frame: 14 days
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 47 | 47 | 46
score on a scale | 6.3 (5.17) | 7.0 (5.60) | 7.0 (6.16)

7. Secondary Outcome: Patient Global Impression for Severity (PGI-S) Global Score
Description: PGI-S us a scale filled by the participant from screening to last visit (all the visits) Participants have to chose 1 condition among 7 : 1 Normal-Not ill at all/ 2 borderline ill/ 3 mildly ill/ 4 moderately ill/ 5 markedly ill/ 6 severely ill/ 7 among the most extremely ill patient
  1 is the best score (very much improved) 7 is the worse score (very much worse)
Time Frame: 14 days
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 47 | 46 | 46
Participants
  normal Not ill at all | 10 | 9 | 8
  borderline ill | 8 | 10 | 10
  mildly ill | 9 | 7 | 9
  moderately ill | 12 | 13 | 11
  markedly ill | 8 | 6 | 5
  severely ill | 0 | 1 | 3

8. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Sleepiness
Description: CGI-C (change from baseline) is a scale completed by the investigator at V3, V4 , V5 and V6 for sleepiness
  the investigator or his/her designee has to score 3 items : global impression/ sleepiness and Cataplexy.
  For each item the investigator or his/her designee has to chose 1 condition among 7 : Very much improved/ Much improved/ Minimally improved/ No change/ Minimally worse/ Much worse/ Very much worse.
  1 is the best score (very much improved) 7 is the worse score (very much worse)
Time Frame: 14 days after the end of treatment period I
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 47 | 47 | 47
Participants
  Very much improved | 6 | 2 | 0
  Much improved | 5 | 11 | 9
  Minimally improved | 16 | 10 | 11
  No change | 14 | 17 | 20
  Minimally worse | 3 | 4 | 6
  Much worse | 3 | 3 | 1
  Very much worse | 0 | 0 | 0

9. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Cataplexy
Description: CGI-C (change from baseline) is a scale completed by the investigator at V3, V4 , V5 and V6 for Cataplexy
  the investigator or his/her designee has to score 3 items : global impression/ sleepiness and Cataplexy.
  For each item the investigator or his/her designee has to chose 1 condition among 7 : Very much improved/ Much improved/ Minimally improved/ No change/ Minimally worse/ Much worse/ Very much worse.
  1 is the best score (very much improved) 7 is the worse score (very much worse)
Time Frame: 14 days after the end of treatment period I
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 40 | 41 | 41
Participants
  Very much improved | 2 | 2 | 0
  Much improved | 1 | 0 | 1
  Minimally improved | 6 | 7 | 7
  No change | 29 | 32 | 33
  Minimally worse | 2 | 0 | 0
  Much worse | 0 | 0 | 0
  very much worse | 0 | 0 | 0

10. Secondary Outcome: Clinical Global Impression for Severity (CGI-S) Global Score
Description: CGI-S is a scale completed by the investigator at each visit : Item global impression
  CGI-S us a scale filled by the Investigator or his/her designee from screening to last visit (all the visits) Investigators have to chose 1 condition among 7 : 1 normal-not ill at all/ 2 borderline ill/ 3 mildly ill/ 4 moderately ill/ 5 markedly ill/ 6 severely ill/ 7 among hte most extremely ill patient
  1 is the best score (very much improved) 7 is the worse score (very much worse)
  CGI-S scale explores 3 items : Global impression/ Sleepiness/ Cataplexy
Time Frame: 14 days after the end of treatment period I
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 48 | 47 | 47
Participants
  normal, not ill at all | 2 | 0 | 1
  borderline ill | 5 | 4 | 7
  mildly ill | 11 | 8 | 11
  moderately ill | 13 | 18 | 14
  markedly ill | 14 | 8 | 5
  severely ill | 3 | 9 | 8
  among the most extremely ill | 0 | 0 | 1

11. Secondary Outcome: Clinical Global Impression for Severity (CGI-S) Sleepiness
Description: CGI-S is a scale completed by the investigator at each visit for Sleepiness
  CGI-S us a scale filled by the Investigator or his/her designee from screening to last visit (all the visits) Investigators have to chose 1 condition among 7 : 1 Normal-Not ill at all/ 2 Borderline ill/ 3 Mildly ill/ 4 Moderately ill/ 5 Markedly ill/ 6 severely ill/ 7 Among the most extremely ill patient
  1 is the best score (very much improved) 7 is the worse score (very much worse)
  CGI-S scale explores 3 items : Global impression/ Sleepiness/ Cataplexy
Time Frame: 14 days after the end of treatment period I
Population: modified Intent To Treat : mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 48 | 47 | 47
Participants
  Normal, not ill at all | 2 | 0 | 1
  Borderline ill | 6 | 3 | 6
  Mildly ill | 9 | 8 | 10
  Moderately ill | 10 | 17 | 12
  Markedly ill | 16 | 10 | 8
  Severely ill | 5 | 9 | 9
  Among the most extremely ill patients | 0 | 0 | 1

12. Secondary Outcome: Clinical Global Impression for Severity (CGI-S) Cataplexy
Description: CGI-S is a scale completed by the investigator at each visit for Cataplexy
  CGI-S us a scale filled by the Investigator or his/her designee from screening to last visit (all the visits) Investigators have to chose 1 condition among 7 : 1 Normal-Not ill at all/ 2 Borderline ill/ 3 Mildly ill/ 4 Moderately ill/ 5 Markedly ill/ 6 severely ill/ 7 Among the most extremely ill patient
  1 is the best score (very much improved) 7 is the worse score (very much worse)
  CGI-S scale explores 3 items : Global impression/ Sleepiness/ Cataplexy
Time Frame: 14 days after the end of treatment period I
Population: modified Intent To Treat : mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 41 | 41 | 41
Participants
  Normal, not ill at all | 7 | 7 | 5
  Borderline ill | 7 | 8 | 14
  Mildly ill | 10 | 10 | 10
  Moderately ill | 10 | 8 | 6
  Markedly ill | 4 | 5 | 0
  Severely ill | 2 | 3 | 6
  Among the most extremely ill patients | 1 | 0 | 0

13. Secondary Outcome: EQ-5D European Quality of Life EQ-5D (Visual Analogic Scale Part)
Description: EQ-5D is a quality of life questionnaire filled in by the participants from screening to the last visit (all visits).
  The EQ-5D is a questionnaire assessing the quality of life of the patient. It has two parts:
  The first part is a descriptive system that assesses five distinct health states/dimensions: Mobility (MO), Self-care (SC), Usual activities (UA), Pain/discomfort, Anxiety/depression (AD). A higher score signifies a higher number of symptoms present.
  The second part is a 100 mm Visual analogic scale (EQ-VAS). An higher score in VAS indicates a better health state.
  The questionnaire is assessed at baseline and all subsequent visits
Time Frame: 14 days
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Modafinil + Placebo | THN102 300/3 | THN102 300/27
Number analyzed (Participants) | 47 | 46 | 46
units on a scale | 70.10 (2.600) | 66.13 (2.601) | 66.72 (2.600)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for each 2 week treatment period during the 3 crossover periods.
Description: Adverse events were collected by investigator - open question to patient. No scale or questionnaire based collection of events.
Groups:
- THN102 300/0: Treatment A : THN102 300/0 Modafinil 300 mg/d Flecainide placebo
  Duration : 2 weeks
- THN102 300/3: Treatment B : THN102 300/3 Modafinil 300 mg/d Flecainide 3 mg/d Duration : 2 weeks
- THN102 300/27: Treatment C : THN102 300/27 Modafinil 300 mg/d Flecainide 27 mg/d Duration : 2 weeks
Arm/Group | THN102 300/0 | THN102 300/3 | THN102 300/27
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 9/48 | 15/47 | 13/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | THN102 300/0 (N=48) | THN102 300/3 (N=47) | THN102 300/27 (N=47)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Palpitation (Cardiac disorders) | 1 | 0 | 0
vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
chalazion (Eye disorders) | 0 | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 1 | 1
dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
toothache (Gastrointestinal disorders) | 1 | 0 | 0
asthenia (General disorders) | 0 | 1 | 0
fatigue (General disorders) | 0 | 0 | 1
hunger (General disorders) | 0 | 0 | 1
sluggishness (General disorders) | 0 | 1 | 0
food allergy (Immune system disorders) | 0 | 0 | 1
gastroenteritis (Infections and infestations) | 0 | 2 | 0
influenza (Infections and infestations) | 0 | 2 | 0
laryngitis (Infections and infestations) | 0 | 1 | 0
nasopharyngitis (Infections and infestations) | 0 | 2 | 2
tracheitis (Infections and infestations) | 0 | 1 | 0
urinary tact infection (Infections and infestations) | 1 | 0 | 0
limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
hepatic enzyme increase (Investigations) | 0 | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
pain in extremity (Metabolism and nutrition disorders) | 0 | 1 | 0
balance disorder (Nervous system disorders) | 1 | 0 | 0
dizziness (Nervous system disorders) | 1 | 0 | 2
dysgeusia (Nervous system disorders) | 0 | 0 | 1
headache (Nervous system disorders) | 2 | 2 | 1
irritability (Psychiatric disorders) | 0 | 1 | 1
nightmare (Psychiatric disorders) | 0 | 1 | 0
violence related symptom (Psychiatric disorders) | 1 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT02821715/SAP_000.pdf
  • Study Protocol (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT02821715/Prot_001.pdf